CLINICAL TRIAL: NCT07005908
Title: Posture and Musculoskeletal System Disorders in Individuals Who Have Had COVID-19
Brief Title: Posture and Pain Measurements in Post-COVID-19
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Associate Professor, Principal Investigator, Izmir Democracy University
Other Study IDs: Effects of COVID on posture
Record Dates: First submitted 2025-06-04; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: COVID-19 Respiratory Infection
Keywords: pain; posture
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-COVID-19 group: This group will consist of individuals who have had COVID-19.
  Interventions: Other: Physical evaluations of post-COVID-19 individuals

INTERVENTIONS:
Other: Physical evaluations of post-COVID-19 individuals — In this study, pain, posture and musculoskeletal disorders were evaluated in post-COVID-19 individuals. The data to be obtained from all these evaluations were collected from the individuals at one time and over a period of approximately 1 hour at the most.

SUMMARY:
In this study, it was aimed to reveal the results of posture measurement evaluated by artificial intelligence method, pain status and musculoskeletal disorders in individuals who have had COVID-19.

DETAILED DESCRIPTION:
Thanks to artificial intelligence and machine learning technology, evaluations such as balance and foot pressure measurement can be made in patients today, as well as applications such as exercise and patient follow-up in rehabilitation, solutions to biomedical problems can be offered. Artificial intelligence and machine learning will continue to play an important role in education, training, patient care and research in the future. On the other hand, although various psychological and physical problems have been shown in individuals who have had COVID-19 during the prolonged COVID-19 pandemic process, musculoskeletal disorders and posture problems in these individuals remain unclear. For this reason, in this study, it was aimed to reveal the results of posture measurement evaluated by artificial intelligence method, pain status and musculoskeletal disorders in individuals who have had COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* adult individuals aged 18 and over
* volunteering to participate in the study,
* Individuals who can understand and answer the questionnaires
* Individuals who were diagnosed with COVID-19 (individuals with a positive Polymerase Chain Reaction (PCR) test result, compatible with COVID-19 infection as a result of lung X-ray or lung tomography despite negative PCR test results) and discharged after recovery/home quarantine completed

Exclusion Criteria:

* Individuals with any physical or mental disability/disease and/or cognitive impairment
* Individuals newly diagnosed with COVID-19, therefore in quarantine at home or receiving treatment in hospital
* Individuals with suspected COVID-19
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 41 individuals with post-COVID-19 were included in the research group.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | through study completion, an average of 1 year
  Pain intensity were measured with the Numerical Rating Scale. This scale expresses the severity of pain with integers from 0 (no pain) to 10 (the worst possible pain).

SECONDARY OUTCOMES:
Posture assessment | through study completion, an average of 1 year
  Posture deviation were determined according to the deviation score in the joint centers obtained by photographing the posture of the individuals and uploading them to the system. Posture assessment were made with a mobile application based on the concept of postural analysis with artificial intelligence.
Score of musculoskeletal disorders | through study completion, an average of 1 year
  The score of musculoskeletal disorders were evaluated using Cornell Musculoskeletal Disorders Questionnaire.A minimum of 0 and a maximum of 90 points are obtained from the scale for each body area. The total score is obtained by adding the scores for each body area. A high total score indicates that the discomfort in the musculoskeletal system is high.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Assoc. Dr., Study Director — Izmir Democracy University; HELİN ÖNCEL, Principal Investigator — Göztepe Sports Club; SİBEL DENİZ, Principal Investigator — Izmir Democracy University; SARA MOHAMMADNEJADIAN, Principal Investigator — Izmir Democracy University; MERVE NUR YÜKSEL, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahuja V, Nair LV. Artificial Intelligence and technology in COVID Era: A narrative review. J Anaesthesiol Clin Pharmacol. 2021 Jan-Mar;37(1):28-34. doi: 10.4103/joacp.JOACP_558_20. Epub 2021 Apr 10. PMID 34103818
- [Background] Itoh N, Mishima H, Yoshida Y, Yoshida M, Oka H, Matsudaira K. Evaluation of the Effect of Patient Education and Strengthening Exercise Therapy Using a Mobile Messaging App on Work Productivity in Japanese Patients With Chronic Low Back Pain: Open-Label, Randomized, Parallel-Group Trial. JMIR Mhealth Uhealth. 2022 May 16;10(5):e35867. doi: 10.2196/35867. PMID 35576560